CLINICAL TRIAL: NCT02093923
Title: A Phase 1b, Double-Blind, Multiple Ascending Dose Study to Assess Safety, Tolerability and Pharmacokinetics of DX-2930 in Hereditary Angioedema Subjects
Brief Title: A Double-Blind, Multiple Ascending Dose Study to Assess Safety, Tolerability and Pharmacokinetics of DX-2930 in Hereditary Angioedema Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DX-2930-02
Record Dates: First submitted 2014-03-17; First posted 2014-03-21 (Estimated); Results first posted 2016-08-01 (Estimated); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Hereditary Angioedema (HAE)
Keywords: HAE
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — lanadelumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- DX-2930, Cohort 1 (Experimental): Participants will receive 30 milligram (mg) dose of DX-2930 subcutaneous (SC) injection once and followed by the second dose after 2 week into the upper arm.
  Interventions: Drug: DX-2930
- DX-2930, Cohort 2 (Experimental): Participants will receive 100 mg dose of DX-2930 SC injection once and followed by the second dose after 2 week into the upper arm.
  Interventions: Drug: DX-2930
- DX-2930, Cohort 3 (Experimental): Participants will receive 300 mg dose of DX-2930 SC injection once and followed by the second dose after 2 week into the upper arm.
  Interventions: Drug: DX-2930
- DX-2930, Cohort 4 (Experimental): Participants will receive 400 mg dose of DX-2930 subcutaneous (SC) injection once and followed by the second dose after 2 week into the upper arm.
  Interventions: Drug: DX-2930
- Placebo (Placebo Comparator): Participants will receive placebo matched to 30, 100, 300 and 400 mg dose of DX-2930 SC injection once and followed by the second dose after 2 week into the upper arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DX-2930 — Participants will receive SC injection of DX-2930 (a recombinant, Chinese hamster ovary [CHO] cell expressed, fully human immunoglobulin IgG1, kappa light chain, monoclonal antibody) once and followed by the second dose after 2 week into the upper arm.
  Arms: DX-2930, Cohort 1; DX-2930, Cohort 2; DX-2930, Cohort 3; DX-2930, Cohort 4
Drug: Placebo — Participants will receive matching placebo subcutaneously.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics (PK) profile of multiple subcutaneous administrations of DX-2930 across a range of doses in HAE participants.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at the time of screening
* Documented diagnosis of HAE (Type I or II)
* Experiencing ≥2 HAE attacks per year, with at least 1 attack in the past 6 months reported by the participant
* Willing and able to read, understand, and sign an informed consent form
* Females of childbearing potential must agree to be abstinent or else use acceptable forms of contraception throughout study
* Males with female partners of childbearing potential must agree to be abstinent or use a medically acceptable form of contraception throughout study

Exclusion Criteria:

* Exposure to an investigational drug or device within 90 days prior to study
* History of exposure within the past 5 years to a monoclonal antibody or recombinant protein bearing an Fc domain
* Concomitant diagnosis of another form of chronic angioedema
* Use of long-term prophylaxis for HAE within 90 days prior to study
* Use of C1-INH that exceeds a total of 30 days within the past 90 days prior to study; any use of C1-INH within 7 days prior to study
* Exposure to angiotensin-converting enzyme (ACE) inhibitors or any estrogen-containing medications with systemic absorption within 90 days prior to study
* Exposure to androgens within 90 days prior to study
* Presence of an indwelling catheter
* Diagnosis of HIV
* Active liver disease or liver function test abnormalities
* History of substance abuse or dependence
* Pregnancy or breastfeeding
* Any condition that, in the opinion of the Investigator, may compromise their safety or compliance, preclude successful conduct of the study, or interfere with interpretation of the results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-05-14 (Actual); Primary Completion 2015-05-18 (Actual); Study Completion 2015-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (14):
- United States (12):
  - UC San Diego Health System - La Jolla, San Diego, California
  - Allergy & Asthma Clinical Research, Walnut Creek, California
  - University of South Florida Asthma, Allergy or Immunology Clinical Research Unit, Tampa, Florida
  - Institute for Asthma & Allergy, PC, Chevy Chase, Maryland
  - Massachusetts General Hospital Allergy Associates, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Winthrop-University Hospital, Clinical Trials Center, Mineola, New York
  - Icahn School of Medicine at Mount Sinai - The Mount Sinai Medical Center, New York, New York
  - UC Physicians Company, Cincinnati, Ohio
  - Baker Allergy, Asthma and Dermatology Research Center, Lake Oswego, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - AARA Research Center, Dallas, Texas
- Ospedale L. Sacco, Milan, MI, Italy
- Jordan University Hospital, Amman, Jordan

REFERENCES:
- [Derived] Banerji A, Busse P, Shennak M, Lumry W, Davis-Lorton M, Wedner HJ, Jacobs J, Baker J, Bernstein JA, Lockey R, Li HH, Craig T, Cicardi M, Riedl M, Al-Ghazawi A, Soo C, Iarrobino R, Sexton DJ, TenHoor C, Kenniston JA, Faucette R, Still JG, Kushner H, Mensah R, Stevens C, Biedenkapp JC, Chyung Y, Adelman B. Inhibiting Plasma Kallikrein for Hereditary Angioedema Prophylaxis. N Engl J Med. 2017 Feb 23;376(8):717-728. doi: 10.1056/NEJMoa1605767. PMID 28225674

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in United States, Italy, and Jordan between 14 May 2014 (first participant first visit) and 18 May 2015 (last participant last visit).
Pre-assignment Details: A total of 38 participants were randomized and 37 participants were treated out of them 36 participants completed the study.
Groups:
- DX-2930, Cohort 1: Participants received 30 milligram (mg) dose of DX-2930 subcutaneous (SC) injection once and followed by the second dose after 2 week into the upper arm.
- DX-2930, Cohort 2: Participants received 100 mg dose of DX-2930 subcutaneous (SC) injection once and followed by the second dose after 2 week into the upper arm.
- DX-2930, Cohort 3: Participants received 300 mg dose of DX-2930 subcutaneous (SC) injection once and followed by the second dose after 2 week into the upper arm.
- DX-2930, Cohort 4: Participants received 400 mg dose of DX-2930 subcutaneous (SC) injection once and followed by the second dose after 2 week into the upper arm.
- Placebo: Participants received placebo matched to 30, 100, 300 and 400 mg dose of DX-2930 subcutaneous (SC) injection once and followed by the second dose after 2 week into the upper arm.
Period: Overall Study
Arm/Group | DX-2930, Cohort 1 | DX-2930, Cohort 2 | DX-2930, Cohort 3 | DX-2930, Cohort 4 | Placebo
Started | 4 | 4 | 5 | 12 | 13
Total Treated | 4 | 4 | 5 | 11 | 13
Treated - 1 Dose Only: | 0 | 0 | 0 | 1 | 0
Treated - 2 Doses: | 4 | 4 | 5 | 10 | 13
Completed | 4 | 4 | 5 | 10 | 13
Not Completed | 0 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0
Not completed — Screen failure after randomization | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population included all randomized participants who received at least 1 dose of study drug.
Groups:
- DX-2930, Cohort 1: Participants received 30 mg dose of DX-2930 subcutaneous (SC) injection once and followed by the second dose after 2 week into the upper arm.
- Total: Total of all reporting groups
Arm/Group | DX-2930, Cohort 1 | DX-2930, Cohort 2 | DX-2930, Cohort 3 | DX-2930, Cohort 4 | Placebo | Total
Number analyzed (Participants) | 4 | 4 | 5 | 11 | 13 | 37
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 5 | 10 | 12 | 35
  >65 years | 0 | 0 | 0 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 1 | 9 | 7 | 23
  Male | 1 | 1 | 4 | 2 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 4 | 4 | 5 | 10 | 13 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 4 | 5 | 11 | 13 | 37
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAE) and Treatment-Emergent Adverse Events (TEAE)
Description: A SAE was any adverse experience occurring at any dose that resulted in any of the following outcomes: Death, Life-threatening experience, required inpatient hospitalization or prolongation of existing hospitalization. Resulted in persistent or significant disability or incapacity. Was a congenital anomaly or birth defect. Was considered to be an important medical event. An AE was considered treatment-emergent if the onset time was after administration of study drug through the Day 120 post-dose final follow-up visit or, in the event that onset time preceded study drug administration, the AE increased in severity during the 120-day post-dose follow-up period.
Time Frame: From Day 1 up to final follow-up (Day 123)
Population: Safety Population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | DX-2930, Cohort 1 | DX-2930, Cohort 2 | DX-2930, Cohort 3 | DX-2930, Cohort 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 5 | 11 | 13
Participants
  Serious Adverse Events | 0 | 0 | 0 | 0 | 1
  Treatment Emergent Adverse Events | 1 | 3 | 2 | 8 | 10

2. Secondary Outcome: Maximum Plasma Concentration (Cmax)
Description: Pharmacokinetic (PK) parameter Cmax data were reported.
Time Frame: Days 1, 2, 4, 8, 15, 16, 18, 22, 29, 36, 50, 64, 92, and 120
Population: Pharmacokinectic (PK) population included all randomized HAE participants in the safety population who had sufficient blood samples to obtain a plasma concentration versus time profile.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | DX-2930, Cohort 1 | DX-2930, Cohort 2 | DX-2930, Cohort 3 | DX-2930, Cohort 4
Number analyzed (Participants) | 4 | 4 | 5 | 9
Nanogram per milliliter (ng/mL) | 3895.0 (2159.76) | 7890.0 (2058.43) | 27460.0 (14542.46) | 45322.2 (8704.56)

3. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax)
Description: PK parameter Tmax data were reported.
Time Frame: Days 1, 2, 4, 8, 15, 16, 18, 22, 29, 36, 50, 64, 92, and 120
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | DX-2930, Cohort 1 | DX-2930, Cohort 2 | DX-2930, Cohort 3 | DX-2930, Cohort 4
Number analyzed (Participants) | 4 | 4 | 5 | 9
Days | 17.930 (1.1400) | 18.020 (0.4596) | 18.172 (1.4526) | 17.700 (0.9804)

4. Secondary Outcome: Area Under the Plasma Concentration-Time Curve (AUC)
Description: PK paramenter AUC data were reported.
Time Frame: Days 1, 2, 4, 8, 15, 16, 18, 22, 29, 36, 50, 64, 92, and 120
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: day*nanogram per milliliter (day*ng/mL)
Arm/Group | DX-2930, Cohort 1 | DX-2930, Cohort 2 | DX-2930, Cohort 3 | DX-2930, Cohort 4
Number analyzed (Participants) | 4 | 4 | 5 | 9
day*nanogram per milliliter (day*ng/mL) | 64100.0 (34731.16) | 135425.0 (48616.76) | 451800.0 (226801.01) | 762777.8 (166713.66)

5. Secondary Outcome: Apparent Clearance (CL/F)
Description: PK parameter CL/F data were reported.
Time Frame: Days 1, 2, 4, 8, 15, 16, 18, 22, 29, 36, 50, 64, 92, and 120
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liter per day (L/day)
Arm/Group | DX-2930, Cohort 1 | DX-2930, Cohort 2 | DX-2930, Cohort 3 | DX-2930, Cohort 4
Number analyzed (Participants) | 4 | 4 | 5 | 9
Liter per day (L/day) | 0.5720 (0.26829) | 0.8110 (0.28258) | 1.0036 (0.90870) | 0.5514 (0.14318)

6. Secondary Outcome: Apparent Volume of Distribution (Vd/F)
Description: PK parameter Vd/F data were reported.
Time Frame: Days 1, 2, 4, 8, 15, 16, 18, 22, 29, 36, 50, 64, 92, and 120
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liter (L)
Arm/Group | DX-2930, Cohort 1 | DX-2930, Cohort 2 | DX-2930, Cohort 3 | DX-2930, Cohort 4
Number analyzed (Participants) | 4 | 4 | 5 | 9
Liter (L) | 11.553 (4.9218) | 16.125 (2.6949) | 17.436 (10.5609) | 11.696 (2.7600)

7. Secondary Outcome: Terminal Elimination Half-Life (t1/2)
Description: PK parameter t(1/2) data were reported.
Time Frame: Days 1, 2, 4, 8, 15, 16, 18, 22, 29, 36, 50, 64, 92, and 120
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | DX-2930, Cohort 1 | DX-2930, Cohort 2 | DX-2930, Cohort 3 | DX-2930, Cohort 4
Number analyzed (Participants) | 4 | 4 | 5 | 9
Day | 14.225 (0.8261) | 14.625 (3.4082) | 13.802 (3.2535) | 14.967 (2.4377)

8. Other Pre Specified Outcome: HAE Attack Rate Per Week From Day 8 to Day 50
Description: Analysis of this outcome measure was based on participants in the 300 mg, 400 mg, and placebo dose groups with a historical baseline attack rate of at least 2 attacks over the last 3 months prior to enrollment. The result is based on General Estimating Equation (GEE) analysis of repeated counts per week during the pre-specified assessment period (Days 8 to 50; predicted to correspond to a period of notable drug exposure). Baseline HAE attack rate per week was a covariate, treatment group is a fixed effect, and participant was a random effect in the GEE model with independence working correlation structure.
Time Frame: Day 8 to Day 50
Population: All randomized participants in the 300 mg, 400 mg, and placebo groups who received at least 1 dose of study drug and who had a historical baseline attack rate of at least 2 attacks in the 3 months prior to enrollment.
Measure: Mean (Standard Error); unit: HAE attacks per week
Groups:
- DX-2930, Combined Cohort 3 and Cohort 4: Participants received 300 mg and 400 mg doses of DX-2930 subcutaneous (SC) injection once and followed by the second dose after 2 week into the upper arm.
- Placebo: Participants received placebo matched to 300 and 400 mg dose of DX-2930 subcutaneous (SC) injection once and followed by the second dose after 2 week into the upper arm.
Arm/Group | DX-2930, Cohort 3 | DX-2930, Cohort 4 | DX-2930, Combined Cohort 3 and Cohort 4 | Placebo
Number analyzed (Participants) | 4 | 11 | 15 | 11
HAE attacks per week
  Mean baseline HAE attack rate (attacks/week) | 0.3269 (0.24627) | 0.5455 (0.17356) | 0.4872 (0.21100) | 0.3916 (0.17694)
  Mean HAE attack rate, unadjusted (attacks/week) | 0 (NA) — No attacks were reported for this arm/group. | 0.0476 (0.15040) | 0.0345 (0.12894) | 0.3636 (0.36376)
  Estimated mean rate based on GEE (attacks/week) | 0 (NA) — No attacks were reported for this arm/group. | 0.0454 (0.03319) | 0.0333 (0.02404) | 0.3712 (0.09596)
Statistical Analysis 1: Comparison: DX-2930, Cohort 3 vs Placebo; The result was based on General Estimating Equation (GEE) analysis. Generalized Estimating Equation (GEE) approach with Poisson distribution assumption was applied to the repeated-measures mixed model with independence working correlation structure. The treatment group was a fixed effect and the number of baseline HAE attacks per week was included as a covariate in the GEE; Test type: Superiority; p < .0001, Mixed Models Analysis; Percent Change in Mean Rate = -100.00, 95% CI 2-sided [-100.00 to -100.00]
Statistical Analysis 2: Comparison: DX-2930, Cohort 4 vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0050, Mixed Models Analysis; Percent Change in Mean Rate = -87.77, 95% CI 2-sided [-97.18 to -46.90]
Statistical Analysis 3: Comparison: DX-2930, Combined Cohort 3 and Cohort 4 vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0012, Mixed Models Analysis; Percent Change in Mean Rate = -91.08, 95% CI [-97.93 to -61.57]

9. Other Pre Specified Outcome: HAE Attacks Per Week From Day 8 to Day 92
Description: This endpoint analysis was based on participants in the 300 mg, 400 mg, and placebo dose groups with a historical baseline attack rate of at least 2 attacks over the last 3 months prior to enrollment. The result is based on General Estimating Equation (GEE) analysis of repeated counts per week during the prespecified assessment period (Day 8 to Day 92 predicted to correspond to a period of notable drug exposure). Baseline HAE attack rate per week is a covariate, treatment group is a fixed effect, and participant is a random effect in the GEE model with independence working correlation structure.
Time Frame: Day 8 to Day 92
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: HAE Attacks per Week
Arm/Group | DX-2930, Cohort 3 | DX-2930, Cohort 4 | DX-2930, Combined Cohort 3 and Cohort 4 | Placebo
Number analyzed (Participants) | 4 | 11 | 15 | 11
HAE Attacks per Week
  Mean baseline HAE attack rate (attacks/week) | 0.3269 (0.24627) | 0.5455 (0.17356) | 0.4872 (0.21100) | 0.3916 (0.17694)
  Mean HAE attack rate, unadjusted (attacks/week) | 0 (NA) — No attacks were reported for this arm/group. | 0.0732 (0.12665) | 0.0526 (0.11206) | 0.3636 (0.36945)
  Estimated mean rate based on GEE (attacks/week) | 0 (NA) — No attacks were reported for this arm/group. | 0.0603 (0.02438) | 0.0461 (0.01826) | 0.3787 (0.10957)
Statistical Analysis 1: Comparison: DX-2930, Cohort 3 vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < .0001, Mixed Models Analysis; Percent Change in Mean Rate = -100.00, 95% CI 2-sided [-100.00 to -100.00]
Statistical Analysis 2: Comparison: DX-2930, Cohort 4 vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < .0001, Mixed Models Analysis; Percent Change in Mean Rate = -84.08, 95% CI 2-sided [-93.07 to -63.46]
Statistical Analysis 3: Comparison: DX-2930, Combined Cohort 3 and Cohort 4 vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < .0001, Mixed Models Analysis; Percent Change in Mean Rate = -87.84, 95% CI 2-sided [-94.81 to -71.50]

10. Other Pre Specified Outcome: HAE Attacks Per Week From Day 8 to Day 64
Description: This endpoint analysis was based on participants in the 300 mg, 400 mg, and placebo dose groups with a historical baseline attack rate of at least 2 attacks over the last 3 months prior to enrollment. The result is based on General Estimating Equation (GEE) analysis of repeated counts per week during the prespecified assessment period (Day 8 to Day 64 predicted to correspond to a period of notable drug exposure). Baseline HAE attack rate per week is a covariate, treatment group is a fixed effect, and participant is a random effect in the GEE model with independence working correlation structure.
Time Frame: Day 8 to Day 64
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: HAE Attacks per Week
Arm/Group | DX-2930, Cohort 3 | DX-2930, Cohort 4 | DX-2930, Combined Cohort 3 and Cohort 4 | Placebo
Number analyzed (Participants) | 4 | 11 | 15 | 11
HAE Attacks per Week
  Mean baseline HAE attack rate | 0.3269 (0.24627) | 0.5455 (0.17356) | 0.4872 (0.21100) | 0.3916 (0.17694)
  Mean HAE attack rate, unadjusted | 0 (NA) — No attacks were reported for this arm/group. | 0.0723 (0.13227) | 0.0522 (0.11651) | 0.3636 (0.33752)
  Estimated mean rate based on GEE | 0 (NA) — No attacks were reported for this arm/group. | 0.0661 (0.02759) | 0.0490 (0.02002) | 0.3773 (0.09518)
Statistical Analysis 1: Comparison: DX-2930, Cohort 3 vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < .0001, Mixed Models Analysis; Percent Change in Mean Rate = -100.00, 95% CI 2-sided [-100.00 to -100.00]
Statistical Analysis 2: Comparison: DX-2930, Cohort 4 vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < .0001, Mixed Models Analysis; Percent Change in Mean Rate = -82.38, 95% CI 2-sided [-92.50 to -58.64]
Statistical Analysis 3: Comparison: DX-2930, Combined Cohort 3 and Cohort 4 vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < .0001, Mixed Models Analysis; Percent Change in Mean Rate = -87.02, 95% CI 2-sided [-94.55 to -69.06]

11. Other Pre Specified Outcome: HAE Attack Rate Per Week From Day 1 to Day 50
Description: This endpoint analysis was based on participants in the 300 mg, 400 mg, and placebo dose groups with a historical baseline attack rate of at least 2 attacks over the last 3 months prior to enrollment. The result is based on General Estimating Equation (GEE) analysis of repeated counts per week during the prespecified assessment period (Day 1 to Day 50 predicted to correspond to a period of notable drug exposure). Baseline HAE attack rate per week is a covariate, treatment group is a fixed effect, and participant is a random effect in the GEE model with independence working correlation structure.
Time Frame: Day 1 to Day 50
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: HAE attacks per week
Arm/Group | DX-2930, Cohort 3 | DX-2930, Cohort 4 | DX-2930, Combined Cohort 3 and Cohort 4 | Placebo
Number analyzed (Participants) | 4 | 11 | 15 | 11
HAE attacks per week
  Mean baseline HAE attack rate (attacks/week) | 0.3269 (0.24627) | 0.5455 (0.17356) | 0.4872 (0.21100) | 0.3916 (0.17694)
  Mean HAE attack rate, unadjusted (attacks/week) | 0 (NA) — No attacks were reported for this arm/group | 0.0541 (0.17634) | 0.0392 (0.15105) | 0.3506 (0.32803)
  Estimated mean rate based on GEE (attacks/week) | 0 (NA) — No attacks were reported for this arm/group. | 0.0525 (0.03998) | 0.0382 (0.02898) | 0.3588 (0.08864)
Statistical Analysis 1: Comparison: DX-2930, Cohort 3 vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < .0001, Mixed Models Analysis; Percent Change in Mean Rate = -100.00, 95% CI 2-sided [-100.00 to -100.00]
Statistical Analysis 2: Comparison: DX-2930, Cohort 4 vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0141, Mixed Models Analysis; Percent Change in Mean Rate = -85.24, 95% CI [-96.79 to -32.03]
Statistical Analysis 3: Comparison: DX-2930, Combined Cohort 3 and Cohort 4 vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0040, Mixed Models Analysis; Percent Change in Mean Rate = -89.35, 95% CI 2-sided [-97.68 to -51.13]

ADVERSE EVENTS:
Time Frame: From Day 1 up to final follow-up (Day 123)
Description: A participant who experienced multiple events within a preferred term was counted once within that preferred term.
Arm/Group | DX-2930, Cohort 1 | DX-2930, Cohort 2 | DX-2930, Cohort 3 | DX-2930, Cohort 4 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/5 | 0/11 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/5 | 0/11 | 1/13
Other Adverse Events (participants affected / at risk) | 1/4 | 3/4 | 2/5 | 8/11 | 10/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DX-2930, Cohort 1 (N=4) | DX-2930, Cohort 2 (N=4) | DX-2930, Cohort 3 (N=5) | DX-2930, Cohort 4 (N=11) | Placebo (N=13)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Pneumonia in both lungs
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DX-2930, Cohort 1 (N=4) | DX-2930, Cohort 2 (N=4) | DX-2930, Cohort 3 (N=5) | DX-2930, Cohort 4 (N=11) | Placebo (N=13)
Hereditary Angioedema (Congenital, familial and genetic disorders) | 0 | 3 | 1 | 5 | 9
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 0 | 1
Injection Site Erythema (General disorders) | 0 | 0 | 0 | 1 | 2
Injection Site Pain (General disorders) | 1 | 2 | 0 | 3 | 3
Pyrexia (General disorders) | 0 | 0 | 0 | 2 | 0
Infleunza (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0
Blood Glucose Increased (Investigations) | 0 | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 2 | 1 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Dyax agreements vary, but Dyax will not prohibit any investigator from publishing. Dyax reviews publications prior to public release and can request deferral by up to 60 days beyond the proposed publication date if necessary to preserve its intellectual property. Dyax can request changes to publications to remove non-study-related confidential information. Dyax can also request deferral of single-center publications until after disclosure of the clinical trial's primary publication.